CLINICAL TRIAL: NCT01309646
Title: Immunogenicity and Safety of GlaxoSmithKline Biologicals' DTPa-IPV/Hib (Infanrix™-IPV+Hib) Vaccine in Healthy Korean Infants
Brief Title: Immunogenicity and Safety of GlaxoSmithKline Biologicals' Infanrix™-IPV+Hib Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 114260; 2012-004137-16 (EudraCT Number)
Record Dates: First submitted 2011-02-24; First posted 2011-03-07 (Estimated); Results first posted 2013-04-02 (Estimated); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Poliomyelitis; Tetanus; Acellular Pertussis; Diphtheria; Haemophilus Influenzae Type b
Keywords: Primary vaccination; combination vaccine; South Korea
MeSH Terms: conditions — Poliomyelitis; Tetanus; Diphtheria; Haemophilus Infections | interventions — Hiberix; PHiD-CV vaccine; RIX4414 vaccine

ARMS (2):
- Infanrix-IPV+Hib Group (Experimental): Subjects aged between, and including, 42 and 69 days at the time of first vaccination received 3 doses of Infanrix™-IPV+Hib at 2, 4 and 6 months of age, 3 doses of Synflorix™ at 6 weeks, 3.5 and 5.5 months of age and 2 doses of Rotarix™ at 6 weeks and 3.5 months of age. The Infanrix™-IPV+Hib was administered intramuscularly in the right thigh, the Synflorix™ vaccine was administered intramuscularly in the left thigh and the Rotarix™ vaccine was administered orally.
  Interventions: Biological: Infanrix™-IPV+Hib; Biological: Synflorix™; Biological: Rotarix™
- Infanrix IPV Group (Active Comparator): Subjects aged between, and including, 42 and 69 days at the time of first vaccination received 3 doses of Infanrix™ IPV and Hiberix™ co-administered at separate injection sites at 2, 4 and 6 months of age, 3 dose of Synflorix™ at 6 weeks, 3.5 and 5.5 months of age and 2 doses of Rotarix™ at 6 weeks and 3.5 months of age. The Infanrix™ IPV was administered intramuscularly in the right thigh, the Synflorix™ and Hiberix™ vaccines were administered intramuscularly in the left thigh and the Rotarix™ vaccine was administered orally.
  Interventions: Biological: Infanrix™ IPV; Biological: Hiberix™; Biological: Synflorix™; Biological: Rotarix™

INTERVENTIONS:
Biological: Infanrix™-IPV+Hib — Intramuscular, 3 doses
  Arms: Infanrix-IPV+Hib Group
Biological: Infanrix™ IPV — Intramuscular, 3 doses
  Arms: Infanrix IPV Group
Biological: Hiberix™ — Intramuscular, 3 doses
  Arms: Infanrix IPV Group
Biological: Synflorix™ — Intramuscular, 3 doses
Biological: Rotarix™ — Oral, 2 doses

SUMMARY:
This study is designed to evaluate the safety and immunogenicity of Infanrix™-IPV+Hib vaccine when administered as a primary vaccination course to healthy Korean infants at 2, 4 and 6 months of age.

ELIGIBILITY:
Inclusion Criteria:

* A male or female between, and including, 42 and 69 days of age at the time of the first vaccination.
* Born after a gestation period of 37 to 42 weeks inclusive.
* Subjects who the investigator believes that parent(s)/Legally Acceptable Representative(s) can and will comply with the requirements of the protocol.
* Written informed consent obtained from the parent(s)/ Legally Acceptable Representative(s) of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Child in care.
* Use of any investigational or non-registered product other than the study vaccine(s) within 30 days preceding the first dose, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs since birth.
* Administration of a vaccine not foreseen by the study protocol, within 30 days prior to the first study visit, with the exception of hepatitis B and Bacillus Calmette-Guérin vaccination; or planned administration during the study period, with the exception of hepatitis B and influenza vaccines, which will be allowed at least 7 days before or 30 days after the administration of the DTPa vaccine.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Evidence of previous or intercurrent diphtheria, tetanus, pertussis, poliomyelitis and Hib vaccination or disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Family history of congenital or hereditary immunodeficiency.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine(s).
* Major congenital defects or serious chronic illness.
* History of any neurological disorders or seizures.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
* Acute disease and/or fever at the time of enrolment.

Ages: 42 Days to 69 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 454 (Actual)
Dates: Start 2011-03-04 (Actual); Primary Completion 2012-02-24 (Actual); Study Completion 2012-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- South Korea (10):
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Goyang
  - GSK Investigational Site, GyeongSangNam-do
  - GSK Investigational Site, Iksan
  - GSK Investigational Site, Jeonju Jeonbuk
  - GSK Investigational Site, Seongnam-si
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon City, Gyeonggi-do
  - GSK Investigational Site, Uijeongbu, Gyeonggi-do
  - GSK Investigational Site, Wonju-si Kangwon-do

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=1691

REFERENCES:
- [Background] Kim KH, Kim CS, Kim HM, Kim JD, Ma SH, Kim DH, Hwang PH, Han JW, Lee TJ, Kim JH, Karkada N, Mesaros N, Sohn WY, Kim JH. Immunogenicity and safety of a combined DTPa-IPV/Hib vaccine administered as a three-dose primary vaccination course in healthy Korean infants: phase III, randomized study. Hum Vaccin Immunother. 2019;15(2):317-326. doi: 10.1080/21645515.2018.1536588. Epub 2018 Nov 15. PMID 30431387

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Initially, a total of 454 subjects were enrolled in the study but 3 subjects had withdrawn from the study. Therefore, a total of 451 subjects were enrolled in the study.
Period: Overall Study
Arm/Group | Infanrix-IPV+Hib Group | Infanrix IPV Group
Started | 224 | 227
Completed | 224 | 227
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Infanrix-IPV+Hib Group | Infanrix IPV Group | Total
Number analyzed (Participants) | 224 | 227 | 451
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 8.8 (1.10) | 8.8 (1.09) | 8.8 (1.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 115 | 212
  Male | 127 | 112 | 239
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - East Asian Heritage | 224 | 226 | 450
  Not specified | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroprotected Subjects for Anti-diphtheria (Anti-D) and Anti-tetanus (Anti-T) Antibodies.
Description: A seroprotected subject was defined as a vaccinated subject who had an anti-D and anti-T antibody concentration equal to or above (≥) 0.1 international units per milliliter (IU/mL).
Time Frame: At Month 5
Population: The analysis was performed on the According-To-Protocol cohort for immunogenicity, which included all evaluable subjects who received one dose of either study vaccine according to their random assignment, for whom administration site of study vaccine was known and for whom immunogenicity data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix-IPV+Hib Group | Infanrix IPV Group
Number analyzed (Participants) | 213 | 217
Participants
  Anti-D | 213 | 217
  Anti-T | 213 | 217

2. Primary Outcome: Number of Seroprotected Subjects for Anti-poliovirus (Anti-polio) Types 1, 2 and 3.
Description: A seroprotected subject was defined as a vaccinated subject who had an anti-polio types 1, 2 and 3 antibody titres equal to or above (≥) 8, cut off corresponding to the effective dose for 50% of the vaccinated subjects.
Time Frame: At Month 5
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix-IPV+Hib Group | Infanrix IPV Group
Number analyzed (Participants) | 212 | 216
Participants
  Anti-Polio 1 | 212 | 216
  Anti-Polio 2: number analyzed (Participants) | 204 | 211
  Anti-Polio 2 | 204 | 211
  Anti-polio 3: number analyzed (Participants) | 198 | 199
  Anti-polio 3 | 197 | 197

3. Primary Outcome: Number of Seroprotected Subjects for Anti-polyribosyl-ribitol-phosphate (Anti-PRP) Antibodies.
Description: A seroprotected subject was defined as a vaccinated subject who had an anti-PRP antibody concentration ≥ 0.15 micrograms per milliliter (µg/mL).
Time Frame: At Month 5
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix-IPV+Hib Group | Infanrix IPV Group
Number analyzed (Participants) | 213 | 217
Participants | 213 | 217

4. Primary Outcome: Anti-pertussis Toxoid (PT), Anti-filamentous Haemagglutinin (FHA) and Anti-pertactin (PRN) Antibody Concentrations.
Description: Concentrations were expressed as geometric mean concentrations (GMCs) for the seropositivity cut-off of 5 ELISA units per milliliter (EL.U/mL).
Time Frame: At Month 5
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Infanrix-IPV+Hib Group | Infanrix IPV Group
Number analyzed (Participants) | 213 | 217
EL.U/mL
  Anti-PT | 54.2 [50.4 to 58.3] | 56 [51.8 to 60.5]
  Anti-FHA | 125 [115.4 to 135.4] | 134.2 [124.2 to 145]
  Anti-PRN | 125.8 [116 to 136.5] | 133.4 [123 to 144.6]

5. Secondary Outcome: Number of Seropositive Subjects for Anti-pertussis Toxoid (PT), Anti-filamentous Haemagglutinin (FHA) and Anti-pertactin (PRN).
Description: A seropositive subjects was defined as a vaccinated subjects who had an anti-PRN, anti-PT and anti-FHA antibody concentration ≥ 5 ELISA units per milliliter (EL.U/mL).
Time Frame: At Month 0 and Month 5
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix-IPV+Hib Group | Infanrix IPV Group
Number analyzed (Participants) | 213 | 217
Participants
  Anti-PT at Month 5 | 213 | 217
  Anti-FHA at Month 5 | 213 | 217
  Anti-PRN at Month 5 | 213 | 217
  Anti-PT at Month 0: number analyzed (Participants) | 212 | 216
  Anti-PT at Month 0 | 27 | 34
  Anti-FHA at Month 0: number analyzed (Participants) | 211 | 214
  Anti-FHA at Month 0 | 170 | 178
  Anti-PRN at Month 0 | 25 | 30

6. Secondary Outcome: Anti-pertussis Toxoid (PT), Anti-filamentous Haemagglutinin (FHA) and Anti-pertactin (PRN) Antibody Concentrations
Description: Concentrations were expressed as geometric mean concentrations (GMCs) for the seropositivity cut-off of 5 EL.U/mL.
Time Frame: At Month 0
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Infanrix-IPV+Hib Group | Infanrix IPV Group
Number analyzed (Participants) | 213 | 217
EL.U/mL
  Anti-PT: number analyzed (Participants) | 212 | 216
  Anti-PT | 3.0 [2.8 to 3.2] | 3.1 [2.9 to 3.3]
  Anti-FHA: number analyzed (Participants) | 211 | 214
  Anti-FHA | 10.5 [9.3 to 12.0] | 11.7 [10.3 to 13.3]
  Anti-PRN | 2.9 [2.7 to 3.0] | 3.1 [2.8 to 3.3]

7. Secondary Outcome: Number of Seroprotected Subjects for Anti-diphtheria (Anti-D) and Anti-tetanus (Anti-T) Antibodies.
Description: as for outcome 1
Time Frame: At Month 0
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix-IPV+Hib Group | Infanrix IPV Group
Number analyzed (Participants) | 213 | 217
Participants
  Anti-D | 29 | 30
  Anti-T | 64 | 76

8. Secondary Outcome: Concentrations for Anti-D and Anti-T Antibodies.
Description: Concentrations were expressed as geometric mean concentrations (GMCs). The seroprotection cut-off of the assay was 0.1 IU/mL.
Time Frame: At Month 0 and Month 5
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Infanrix-IPV+Hib Group | Infanrix IPV Group
Number analyzed (Participants) | 213 | 217
IU/mL
  Anti-D at Month 0 | 0.058 [0.055 to 0.061] | 0.060 [0.056 to 0.064]
  Anti-D at Month 5 | 8.096 [7.520 to 8.717] | 8.692 [8.125 to 9.298]
  Anti-T at Month 0 | 0.081 [0.072 to 0.090] | 0.091 [0.080 to 0.103]
  Anti-T at Month 5 | 10.259 [9.654 to 10.902] | 12.421 [11.599 to 13.301]

9. Secondary Outcome: Number of Seroprotected Subjects Anti-poliovirus (Anti-polio) Types 1, 2 and 3.
Description: as for outcome 2
Time Frame: At Month 0
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix-IPV+Hib Group | Infanrix IPV Group
Number analyzed (Participants) | 211 | 216
Participants
  Anti-Polio 1 | 104 | 89
  Anti-Polio 2: number analyzed (Participants) | 211 | 214
  Anti-Polio 2 | 119 | 108
  Anti-polio 3 | 41 | 31

10. Secondary Outcome: Titres for Anti-polio Types 1, 2 and 3.
Description: Titres were expressed as geometric mean titres (GMTs). The seroprotection cut-off of the assay was 8.
Time Frame: At Month 0 and Month 5
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Infanrix-IPV+Hib Group | Infanrix IPV Group
Number analyzed (Participants) | 212 | 216
titers
  Anti-polio 1 at Month 0: number analyzed (Participants) | 211 | 216
  Anti-polio 1 at Month 0 | 9.5 [8.3 to 11.0] | 9.4 [8.0 to 11.0]
  Anti-polio 1 at Month 5 | 328.8 [289.8 to 373.1] | 372.7 [323.8 to 428.9]
  Anti-polio 2 at Month 0: number analyzed (Participants) | 211 | 214
  Anti-polio 2 at Month 0 | 10.8 [9.4 to 12.5] | 8.8 [7.7 to 9.9]
  Anti-polio 2 at Month 5: number analyzed (Participants) | 204 | 211
  Anti-polio 2 at Month 5 | 340.6 [295.4 to 392.6] | 400.2 [347.6 to 460.7]
  Anti-polio 3 at Month 0: number analyzed (Participants) | 211 | 216
  Anti-polio 3 at Month 0 | 5.5 [5.0 to 6.1] | 4.9 [4.5 to 5.3]
  Anti-polio 3 at Month 5: number analyzed (Participants) | 198 | 199
  Anti-polio 3 at Month 5 | 377.7 [322.3 to 442.6] | 465.3 [390.3 to 554.7]

11. Secondary Outcome: Number of Seroprotected Subjects for Anti-polyribosyl-ribitol-phosphate (Anti-PRP) Antibodies.
Description: as for outcome 3
Time Frame: At Month 0
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix-IPV+Hib Group | Infanrix IPV Group
Number analyzed (Participants) | 213 | 217
Participants | 91 | 109

12. Secondary Outcome: Concentrations of Anti-PRP Antibodies.
Description: Concentrations were expressed as geometric mean concentrations (GMCs). The seroprotection cut-off of the assay was 0.15 µg/mL.
Time Frame: At Month 0 and Month 5
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Infanrix-IPV+Hib Group | Infanrix IPV Group
Number analyzed (Participants) | 213 | 217
µg/mL
  Anti-PRP at Month 0 | 0.165 [0.143 to 0.191] | 0.219 [0.184 to 0.260]
  Anti-PRP at Month 5 | 8.456 [7.283 to 9.819] | 18.700 [16.353 to 21.384]

13. Secondary Outcome: Number of Subjects With a Vaccine Response to Anti-PT, Anti-FHA and Anti-PRN.
Description: Vaccine response was defined as antibody concentration ≥ 5 EL.U/mL at post vaccination, for initially seronegative subjects, and at least maintenance of antibody concentration from pre to post-vaccination (i.e. antibody concentration at post vaccination ≥ 1 fold the pre-vaccination antibody concentration), for initially seropositive subjects.
Time Frame: At Month 5
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix-IPV+Hib Group | Infanrix IPV Group
Number analyzed (Participants) | 213 | 217
Participants
  Anti-PT: number analyzed (Participants) | 212 | 216
  Anti-PT | 211 | 215
  Anti-FHA: number analyzed (Participants) | 211 | 214
  Anti-FHA | 207 | 207
  Anti-PRN | 213 | 216

14. Secondary Outcome: Number of Subjects With Any Solicited Local Symptoms.
Description: Assessed solicited local symptoms were pain, redness and swelling at the injection site. Any = incidence of a particular symptom regardless of intensity grade.
Time Frame: During the 4-day (Days 0-3) follow-up period after any vaccination with Infanrix™-IPV+Hib or Infanrix™ IPV + Hiberix™
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one vaccine administration documented and with the symptom sheet completed.
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix-IPV+Hib Group | Infanrix IPV Group
Number analyzed (Participants) | 224 | 227
Participants
  Any Pain | 143 | 146
  Any Redness | 177 | 167
  Any Swelling | 130 | 121

15. Secondary Outcome: Number of Subjects With Any Solicited General Symptoms.
Description: Assessed solicited general symptoms were drowsiness, irritability/fussiness, loss of appetite and fever [defined as tympanic temperature ≥ 37.5 degrees Celsius (°C)]. Any = incidence of a particular symptom regardless of intensity grade.
Time Frame: During the 4-day (Days 0-3) follow-up period after any vaccination with Infanrix™-IPV+Hib or Infanrix™ IPV + Hiberix™
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix-IPV+Hib Group | Infanrix IPV Group
Number analyzed (Participants) | 224 | 227
Participants
  Any Drowsiness | 153 | 147
  Any Irritability/Fussiness | 181 | 182
  Any Loss of appetite | 120 | 103
  Temperature ≥ 37.5°C | 83 | 81

16. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs).
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any = any unsolicited AE regardless of intensity or relationship to vaccination.
Time Frame: During the 31-day (Days 0-30) follow-up period after any vaccination with Infanrix™-IPV+Hib or Infanrix™ IPV + Hiberix™
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix-IPV+Hib Group | Infanrix IPV Group
Number analyzed (Participants) | 224 | 227
Participants | 130 | 123

17. Secondary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs).
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period (from Month 0 to Month 7)
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix-IPV+Hib Group | Infanrix IPV Group
Number analyzed (Participants) | 224 | 227
Participants | 25 | 21

ADVERSE EVENTS:
Time Frame: SAE(s): during the entire study period (Month 0 to Month 7); Solicited local/general symptoms: during the 4-day (Days 0-3) follow-up period after any vaccination; Unsolicited AE(s): during the 31-day (Days 0-30) follow-up period after any vaccination.
Arm/Group | Infanrix-IPV+Hib Group | Infanrix IPV Group
All-Cause Mortality (participants affected / at risk) | 0/224 | 0/227
Serious Adverse Events (participants affected / at risk) | 25/224 | 21/227
Other Adverse Events (participants affected / at risk) | 218/224 | 220/227
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infanrix-IPV+Hib Group (N=224) | Infanrix IPV Group (N=227)
Bronchiolitis (Infections and infestations) | 7 | 5
Urinary tract infection (Infections and infestations) | 1 | 6
Pneumonia (Infections and infestations) | 5 | 1
Gastroenteritis (Infections and infestations) | 4 | 1
Viral infection (Infections and infestations) | 1 | 3
Bronchitis (Infections and infestations) | 2 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 1
Pharyngitis (Infections and infestations) | 2 | 0
Skull fracture (Injury, poisoning and procedural complications) | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Croup infectious (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Intussusception (Gastrointestinal disorders) | 1 | 0
Meningitis (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Pyelonephritis chronic (Infections and infestations) | 0 | 1
Respiratory syncytial virus bronchitis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Vesicoureteric reflux (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Infanrix-IPV+Hib Group (N=224) | Infanrix IPV Group (N=227)
Nasopharyngitis (Infections and infestations) | 37 | 29
Upper respiratory tract infection (Infections and infestations) | 34 | 29
Diarrhoea (Gastrointestinal disorders) | 29 | 10
Bronchitis (Infections and infestations) | 14 | 14
Bronchiolitis (Infections and infestations) | 14 | 13
Pain (General disorders) | 143 | 146
Redness (General disorders) | 177 | 167
Swelling (General disorders) | 130 | 121
Drowsiness (General disorders) | 153 | 147
Irritability/Fussiness (General disorders) | 181 | 182
Loss of appetite (General disorders) | 120 | 103
Temperature (Tympanic) (General disorders) | 83 | 81

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.